CLINICAL TRIAL: NCT04471064
Title: A Multicenter, Open, Dose Increasing Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Primary Efficacy of xy0206 Tablets in Relapsed / Refractory Acute Myeloid Leukemia Subjects
Brief Title: A Study of XY0206 Tablets in Patients With Relapsed / Refractory Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shijiazhuang Yiling Pharmaceutical Co. Ltd (Industry)
Collaborators: Proswell Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HY-XY0206-Ⅰ-02
Record Dates: First submitted 2020-07-01; First posted 2020-07-14 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- XY0206-12.5mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：12.5mg; multiple dose phase
  Interventions: Drug: XY0206
- XY0206-25mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：25mg; multiple dose phase
  Interventions: Drug: XY0206
- XY0206-50mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：50mg; multiple dose phase
  Interventions: Drug: XY0206
- XY0206-100mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：100mg; multiple dose phase
  Interventions: Drug: XY0206
- XY0206-150mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：150mg; multiple dose phase
  Interventions: Drug: XY0206
- XY0206-200mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：200mg; multiple dose phase
  Interventions: Drug: XY0206
- XY0206-250mg (Experimental): Drug:XY0206;Dosage form:Tablet;Dosage：250mg; multiple dose phase
  Interventions: Drug: XY0206

INTERVENTIONS:
Drug: XY0206 — Dosage form:Tablet;Multiple dose phase:Take the medicine once a day,1 tablet at a time.4 weeks of continuous medication is one course of treatment. After the first course of treatment, the subjects can continue to receive the experimental drug treatment until they meet the withdrawal criteria. The duration and interval of treatment were determined according to the accumulated condition after multiple dose.

SUMMARY:
1. To evaluate the safety and tolerability of xy0206 as single drug in the treatment of relapsed / refractory AML;
2. Evaluate the dose limited toxicity (DLT) and maximum tolerable dose (MTD) of xy0206 as single drug in the treatment of relapsed / refractory AML subjects.
3. To evaluate the pharmacokinetic (PK), pharmacokinetic (PD) characteristics and PK / PD correlation of xy0206 as single drug treatment in relapsed / refractory AML subjects;
4. To evaluate the primary efficacy of xy0206 as single drug in the treatment of relapsed / refractory AML patients;
5. To evaluate biomarkers of xy0206 as single drug treatment for relapsed / refractory AML subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patients must meet all of the following criteria before entering the group:

  1. At least 18 years old; 2. Based on the World Health Organization (WHO) 2016 classification, the patients who were confirmed by the morphology of bone marrow cells and met the diagnosis criteria of relapsed / refractory AML (refer to the Chinese diagnosis and treatment guidelines for relapsed and refractory acute myeloid leukemia (2017 version)), the diagnosis criteria of relapsed AML: after CR, the peripheral blood once again showed leukemia cells or the original / immature cells in bone marrow were more than 5% (except the bone marrow after consolidated chemotherapy) The diagnosis standard of refractory AML: the primary refractory disease that has not been completely relieved after two courses of chemotherapy induced by standard regimen (including cytarabine and an anthracycline or anthraquinone drug); 3. ECOG physical fitness score is ≤ 2 points ; 4 Estimated survival time ≥ 12 weeks; 5 The organ function level of subjects must meet the following requirements:
  * Blood routine test: WBC ≤ 30 × 109 / L (it is allowed to take hydroxyurea until 3 days before administration of test drug to stabilize WBC);
  * Blood biochemistry: serum creatinine (Scr) ≤ 1.5 × ULN or creatinine clearance rate (Ccr) ≥ 60 ml / min (using Cockcroft -Gault formula); alanine aminotransferase (ALT), aspartate aminotransferase (AST) and alkaline phosphatase (ALP) ≤ 2.5 × ULN (liver with leukemia cell infiltration ≤ 5 × ULN), total bilirubin (TBIL) ≤ 1.5 × ULN;
  * Electrolyte: the content of potassium, sodium, calcium and magnesium in the blood is within the normal value range of the laboratory (if the abnormal laboratory result judged by the researcher is of no clinical significance or can be controlled within the normal value range by drugs in the screening period, the subject can be included in the group);
  * Coagulation function: INR ≤ 1.5 × ULN, APTT < 10 seconds, PT < 3 seconds, FIB ≥ 1.5g/l (blood products or drugs are allowed to be corrected 3 days before administration of test drugs);
  * Friderica corrected QT value (QTC) for male ≤ 450 ms or female ≤ 470 MS;
  * LVEF≥ 50%；
  * Urinary protein < 2 + was detected in urine routine. If urinary protein ≥ 2 +, 24-hour urinary protein quantification is needed, and only when 24-hour urinary protein < 2g can be enrolled in the group; 6. The serum pregnancy test must be carried out within 28 days before receiving the first dose of study drug and the result must be negative. The women of childbearing age and the male subjects agree to adopt the routine and effective contraceptive measures during the whole study period and within 6 months after the treatment; 7. The subjects should be willing to provide effective diagnosis evidence before treatment or accept bone marrow puncture or biopsy for diagnosis, and accept bone marrow puncture or biopsy for efficacy evaluation after treatment; 8. Volunteer to participate in clinical research and sign informed consent in writing.

Exclusion Criteria:

* Patients cannot participate in this clinical study if they meet any of the following conditions:

  1. Known allergy to the study drug or any of its ingredients; has been treated with sunitinib malate, or allergy to sunitinib malate;
  2. BCR / ABL positive leukemia (chronic myeloid leukemia);
  3. The subjects had central nervous system leukemia;
  4. The subjects had secondary AML after chemotherapy for other tumors (except MDS);
  5. At the same time, patients with other malignant tumors (except for those with cured stage IB or lower grade cervical cancer, non-invasive basal cell or squamous cell skin cancer, malignant melanoma with complete remission (CR) > 10 years, and other malignant tumors with complete remission (CR) > 5 years);
  6. Treatment before the trial:

     * Previous treatment with FLT3 inhibitor;
     * Patients who have received allogeneic hematopoietic stem cell transplantation before;
     * Received chemotherapy, biotherapy, targeted antitumor therapy within 28 days before starting to use the study drug, and radiotherapy within 14 days;
     * Drugs with significant effect on P450 metabolic enzyme pathway taken within 2 weeks before the screening period;
     * Have participated in other clinical studies and applied research drugs within 28 days before starting to use research drugs;
     * Major surgery or significant traumatic injury within 28 days prior to the first administration of the study treatment or maybe major surgery is needed during the study treatment period;
     * Concomitant drugs that may cause QTc prolongation or induce torsade de pointes (TdP) are required, in addition to antimicrobials used as standard therapy for the prevention or treatment of infection and other such drugs considered essential by the researchers;
  7. The toxic and side effects caused by previous treatment did not recover to CTCAE ≤ 1, except for hair loss and other tolerable events judged by the researchers;
  8. Combined diseases:

     * One or more HBsAg, HCV, anti HIV or anti Treponema pallidum specific antibodies are positive;
     * Clinically significant gastrointestinal abnormalities that may affect drug intake, transport or absorption (e.g., inability to swallow, chronic diarrhea, intestinal obstruction, peptic ulcer, etc.), subjects with total gastrectomy, or patients with malabsorption syndrome;
     * Have a history of uncontrolled epilepsy, central nervous system disease or mental illness;
     * Hypertension with poor drug control (persistent systolic blood pressure ≥ 150 mmHg and / or diastolic blood pressure ≥ 100 mmHg despite antihypertensive treatment);
     * Poorly controlled diabetes mellitus (fasting blood glucose continues to be > 7.1mmol/L despite hypoglycemic treatment), or insulin-dependent diabetes mellitus (type I diabetes), or non insulin-dependent diabetes mellitus with small vessel disease, or pancreatic dysfunction;
     * In the 12 months before the first application, there were any of the following conditions: symptomatic congestive heart failure (New York Heart Association class II-IV), uncontrolled arrhythmia, angina pectoris, myocardial infarction, stroke (except lacunar infarction), coronary / peripheral artery bypass surgery, pulmonary embolism;
     * Long QT syndrome with congenital long QT interval syndrome or known family history;
     * There is a history of LVEF falling below 40%;
     * Uncontrolled active infections (bacteria, viruses, fungi, etc.);
     * Bleeding grade ≥ grade 3 ;
     * Have adrenal insufficiency;
     * The thyroid function was abnormal in the past, or could not be maintained in the normal range even under the condition of drug treatment;
     * Currently, there are serious unhealed wounds, ulcers or fractures;
     * Stevens Johnson syndrome (SJS) and toxic epidermal necrolysis (TEN);
  9. For female subjects: currently in pregnancy or lactation;
  10. Any previous or current disease, treatment, or laboratory abnormality that may interfere with the results of the study, affect the subject's participation in the whole process of the study, or the subject is not suitable for the study in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerable dose | from the start of the medication to the end of the study or 28 days after cessation of medication
  The occurrence of Maximum tolerable dose.
Dose limiting toxicity | from the start of the medication to the end of the study or 28 days after cessation of medication
  The occurrence of Dose limiting toxicity.
Adverse event | from the start of the medication to the end of the study or 28 days after cessation of medication
  The occurrence rate of Adverse event.
Adverse drug reactions | from the start of the medication to the end of the study or 28 days after cessation of medication
  The occurrence rate of adverse drug reactions.
Serious adverse events | from the start of the medication to the end of the study or 28 days after cessation of medication
  The occurrence rate of Serious adverse events.
Blood routine | from the start of the medication to the end of the study or 28 days after cessation of medication
  Check whether the red blood cell system, white blood cell system and platelet system are normal
Urine routine | from the start of the medication to the end of the study or 28 days after cessation of medication
  Urine routine examination includes urine color, transparency, pH, red blood cells, white blood cells, epithelial cells, tube type, protein, specific gravity and urine sugar.
Stool routine | from the start of the medication to the end of the study or 28 days after cessation of medication
  Routine stool tests include the detection of red and white blood cells in feces, bacterial sensitivity test, occult blood test (OB) and inspection of eggs.
Blood biochemistry | from the start of the medication to the end of the study or 28 days after cessation of medication
  The contents of various ions, sugars, lipids, proteins, enzymes, hormones and metabolites in blood were detected
Serum amylase / lipase | from the start of the medication to the end of the study or 28 days after cessation of medication
  Evaluation of pancreatic function
Coagulation function | from the start of the medication to the end of the study or 28 days after cessation of medication
  Four coagulation parameters including prothrombin time (PT), activated partial thromboplastin time (APTT), thrombin time (TT) and fibrinogen (FIB) were evaluated.
ECG | from the start of the medication to the end of the study or 28 days after cessation of medication
  Evaluation of QT interval
Echocardiography | from the start of the medication to the end of the study or 28 days after cessation of medication
  To evaluate the electrophysiological condition of the heart
Imaging examination | from the start of the medication to the end of the study or 28 days after cessation of medication
  Chest X-ray/CT
Body temperature | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the vital signs.
Blood pressure | from the start of the medication to the end of the study or 28 days after cessation of medication
  Assess whether systolic blood pressure and diastolic blood pressure are normal
Heart rate | from the start of the medication to the end of the study or 28 days after cessation of medication
  One of the vital signs.
Breathing | from the start of the medication to the end of the study or 28 days after cessation of medication
  Assess if breathing is normal
Skin | from the start of the medication to the end of the study or 28 days after cessation of medication
  Assess if the skin is normal.
Head | from the start of the medication to the end of the study or 28 days after cessation of medication
  Head examination includes head, eyes, ears, nose, lips, etc.Assess if head is normal
Neck | from the start of the medication to the end of the study or 28 days after cessation of medication
  Neck examination includes thyroid gland, lymph node, etc.Assess if neck is normal.
Chest | from the start of the medication to the end of the study or 28 days after cessation of medication
  Chest examination includes lung, cardiovascular, etc.Assess if chest is normal.
Abdomen | from the start of the medication to the end of the study or 28 days after cessation of medication
  Abdominal examination includes liver and spleen.Assess if abdomen is normal.
Limbs | from the start of the medication to the end of the study or 28 days after cessation of medication
  Assess if limbs is normal.
Nerves | from the start of the medication to the end of the study or 28 days after cessation of medication
  Assess nerve function by communication
Back/spine | from the start of the medication to the end of the study or 28 days after cessation of medication
  Assess if back/spine is normal.

CONTACTS AND LOCATIONS:
Overall Officials: Junyuan Qi, MD, Principal Investigator — Institute of Hematology, Chinese Academy of Medical Sciences
Locations (1):
- Institute of Hematology, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No